CLINICAL TRIAL: NCT05966116
Title: Sodium Accumulation Study in Haemodialysis: Brain Study
Acronym: SASH-B
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2023/055
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Dialysis; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the research study is to look at a new type of MRI scanning that can measure the amount of sodium in different parts of the body. Sodium (or 'salt') levels are very important in maintaining health, and high levels lead to high blood pressure. This is very important to patients with kidney disease, as the kidney is the main organ that regulates the amount of sodium in the body. It is possible to measure blood sodium levels, but this does not tell us how much sodium is present in other areas of the body. Previously, it has not been possible measure this. Sodium MRI (Na-MRI) is a new type of MRI scanning that can directly measure sodium in other parts of body such as skin, muscles, kidneys, and brain. The investigators believe that this will help to guide treatment in patients with kidney disease who are on haemodialysis, research studies are needed to prove the benefits.

DETAILED DESCRIPTION:
Haemodialysis (HD) sustains life in patients with end-stage kidney disease (ESKD) but is associated with a marked increase in cognitive impairment, being three times more common and presenting at a younger age. The predominant features of cognitive impairment associated with HD are loss of executive function, including higher processing such as planning, task prioritisation and self-regulation. The mechanism for development and acceleration of cognitive impairment on dialysis is not well understood, however hypertension and cardiovascular disease are likely to play a significant role, alongside changes in brain perfusion as a result of dialysis itself, which has been shown in a prior study using PET-CT.

Sodium balance is normally regulated by the kidneys in health, but has to be achieved by sodium removal during HD for those with ESKD. Recent evidence suggests that accumulation of sodium in tissue may be a critical factor impacting the development of hypertension and cardiovascular disease (CVD) in patients with ESKD. Non-invasive methods are therefore required to study tissue sodium accumulation in this context.

23Na MRI has the potential to provide complementary quantitative parameters of tissue health, in a non-invasive manner. Sodium homeostasis is central to maintenance of human physiology, providing an index of cellular integrity and energy status. The maintenance of sodium gradients across the cell membrane, by the Na+/K+ ATPase pump, enables 23Na MRI to distinguish between different environments within organs, providing a biomarker of disease status, notably kidney disease, hypertension, and brain disorders.

Previously, traditional proton (1H) magnetic resonance imaging (MRI) in dialysis patients demonstrated a decrease in grey matter T1 and an accompanying increase in white matter T1 when comparing scans before, during and after dialysis, In this context, T1 can be thought of as a marker of water content. This demonstrates that changes in the brain occur as a direct consequence of dialysis, with fluid and sodium shifts across cellular compartments the most likely explanation. This is important, as it suggests a novel mechanism by which dialysis may cause reductions in cognitive function. However, this needs further study to establish these mechanisms with more confidence.

At the SPMIC, a dual tuned proton(1H)/sodium(23Na) volume head RF coil for 23Na imaging of the brain has been installed and interfaced; and imaging methods to perform 23Na MRI of the brain have been optimised.

This study proposes to utilise 23Na MRI of the brain along with proton measures of T1, before and after dialysis within existing experimental set-up at SPMIC. This will provide new insights into the direct effects of dialysis on brain sodium levels, and in turn deepen our understanding of the link between sodium, fluid overload, dialysis and the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years inclusive
* Male and female patients with CKD stage 5 receiving chronic haemodialysis
* Patient has been dialysis dependent for at least 3 months
* Must be able to follow simple instruction in English (on safety ground for MRI scans) and be able to understand the nature and requirements of the study

Exclusion Criteria:

* Active infection or malignancy
* Amputee
* Pregnancy
* Contraindication to MRI scanning including claustrophobia, pacemaker, metallic implants etc
* Unable or unwilling to provide informed consent
* Medical conditions or overall physical frailty precludes scan session in opinion of investigator
* Any condition which could interfere with the patient's ability to comply with the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 participants (5 male and 5 female) who are over 50 and under 75 years old who have been on haemodialysis for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of brain images that can be analysed for sodium levels | 12 months
  success criterion > 85%

SECONDARY OUTCOMES:
Change in grey and white matter sodium levels | 12 months
  comparing before and after dialysis
Association between change in brain sodium levels to proton MRI measures | 12 months
  grey/white matter volume, T1

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Noble, BMBS, Principal Investigator — The University of Nottingham
Locations (1):
- Centre for Kidney Research and Innovation, Derby, United Kingdom